CLINICAL TRIAL: NCT02278471
Title: The SCCS Polypill Pilot Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Thomas Wang, Director of the Division of Cardiovascular Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 141583
Record Dates: First submitted 2014-10-13; First posted 2014-10-30 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Hypertension; Hyperlipidemia
Keywords: combination pill; polypill; primary prevention
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Atorvastatin; Amlodipine; Losartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Subjects in this arm will not receive any investigational medications. They will remain on the same care that they are use to receiving.
- Polypill (Experimental): The study medication will be a fixed-dose combination pill (polypill) containing: Atorvastatin 10 mg, amlodipine 2.5 mg, losartan 25 mg, and hydrochlorothiazide 12.5 mg.
  Polypill will be taken once daily.
  Interventions: Drug: Polypill (atorvastatin, amlodipine, losartan, and hydrochlorothiazide)

INTERVENTIONS:
Drug: Polypill (atorvastatin, amlodipine, losartan, and hydrochlorothiazide)
  Arms: Polypill

SUMMARY:
In this study the investigators will examine the effect of the polypill on medication adherence, systolic blood pressure, and LDL cholesterol over a 12 month span.

DETAILED DESCRIPTION:
The purpose of this study is to assess if a polypill-based approach to primary CVD prevention is feasible in a low socioeconomic status population. The study will assess whether a polypill approach is associated with better cardiovascular risk factor control compared with usual care.

The polypill will be supplied as a compounded pill containing atorvastatin 10 mg, amlodipine 2.5 mg, losartan 25 mg, and hydrochlorothiazide 12.5 mg. The medications in the polypill have been extensively evaluated individually and in combination. Each of the medications in the polypill is approved by the United States Food and Drug Administration (FDA) and widely administered in the US for the treatment of and prevention of cardiovascular disease. The doses of each component medication included in the polypill are low, which should minimize the chance of any potential side-effects.

In this study we assess medication adherence, systolic blood pressure, and LDL cholesterol over a 12 month span, in subjects taking the polypill versus subjects under usual care.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at the SCCS site in Mobile, Alabama, obtain care at Franklin Primary Health Center, or live in the surrounding area.
* Aged 45-75 years
* Baseline systolic blood pressure ≥120 mm Hg. In this open-label trial, the study physicians are permitted to prescribe any additional medication deemed appropriate to achieve blood pressure control.

Exclusion Criteria:

* History of coronary heart disease or stroke
* History of cancer, except for basal cell skin cancer
* History of liver disease, not including chronic, clinically-stable hepatitis
* Laboratory evidence of hepatic dysfunction (an alanine aminotransferase level more than two times the upper limit of the normal range)
* Known renal disease, estimated creatinine clearance < 60
* Current use of more than 2 anti-hypertensive medications
* LDL cholesterol ≥190 mg/dl
* Insulin-dependent diabetes
* Known intolerance to any of the components of the polypill
* Potassium <3.4 or >5.5 mEq/L
* Use of medications that interact with statins, including those affecting the cytochrome P450 system
* Current use of diuretics for indications other than hypertension
* Comorbidities that might be expected to limit lifespan during the 12-month follow-up period
* Inability to provide consent.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Wang, MD, Principal Investigator — Vanderbilt Univeristy
Locations (1):
- Franklin Primary Health Center, Mobile, Alabama, United States

REFERENCES:
- [Derived] Munoz D, Uzoije P, Reynolds C, Miller R, Walkley D, Pappalardo S, Tousey P, Munro H, Gonzales H, Song W, White C, Blot WJ, Wang TJ. Polypill for Cardiovascular Disease Prevention in an Underserved Population. N Engl J Med. 2019 Sep 19;381(12):1114-1123. doi: 10.1056/NEJMoa1815359. PMID 31532959

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Potentially eligible participants were invited to complete a baseline visit. During baseline visit, if eligibility confirmed, patients then randomized in open-label 1:1 fashion to either polypill arm or usual care arm. Only if baseline visit labs yielded an exclusionary result were participants then disqualified from further study participation.
Groups:
- Usual Care: Subjects in this arm will not receive any investigational medications. They will continue to receive usual medical care, as directed by their primary care providers.
- Polypill: The study medication will be a fixed-dose combination pill (polypill) containing: Atorvastatin 10 mg, amlodipine 2.5 mg, losartan 25 mg, and hydrochlorothiazide 12.5 mg.
  Polypill will be taken once daily.
  Polypill (atorvastatin, amlodipine, losartan, and hydrochlorothiazide)
Period: Overall Study
Arm/Group | Usual Care | Polypill
Started | 155 | 148
Completed | 147 | 128
Not Completed | 8 | 20
Not completed — Lost to Follow-up | 6 | 15
Not completed — Death | 2 | 2
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Polypill | Total
Number analyzed (Participants) | 155 | 148 | 303
Age, Continuous [Median (Standard Deviation); unit: years] — Mean age was the same for both the Polypill and the Usual care arms.
  years | 56 (6) | 56 (6) | 56 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 65 | 164
  Male | 56 | 83 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 151 | 141 | 292
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 155 | 148 | 303
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 140 (17) | 140 (18) | 140 (17)
LDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 112 (37) | 114 (32) | 113 (34)

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: polypill versus usual care
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Usual Care | Polypill
Number analyzed (Participants) | 147 | 128
mm Hg | 138 (23) | 131 (21)

2. Primary Outcome: Medication Adherence-Percentage of Pills Taken
Description: polypill arm-evaluation via pill counts.
Time Frame: 12 months
Population: adherence not assessed in usual care arm; incomplete data for 27 polypill participants, resulting in 101 analyzed of 128 polypill participants who completed 12 month visits
Measure: Median (Inter-Quartile Range); unit: percentage of pills taken
Arm/Group | Usual Care | Polypill
Number analyzed (Participants) | 0 | 101
percentage of pills taken |  | 86 [79 to 93]

3. Primary Outcome: LDL Cholesterol
Description: Polypill versus usual care
Time Frame: 12 months
Population: # of participants in polypill arm analyzed (126) does not match number of polypill participants completed (128; in the participant flow overview) because we were unable to obtain LDL values at baseline for 2 Polypill participants. The lab was unable to calculate and a reflex direct LDL was not processed.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | Polypill
Number analyzed (Participants) | 147 | 126
mg/dL | 109 (32) | 98 (35)

4. Secondary Outcome: Systolic Blood Pressure
Description: polypill versus usual care
Time Frame: 2 months
Population: The numbers of participants analyzed do not match those of the completed (in the participant flow overview) because this assessment was completed at baseline and 2 months; 291 patients (153 usual care, 138 Polypill) completed 2-month follow-up, whereas 275 (147 Usual Care, 128 Polypill) completed 12-month follow-up.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Usual Care | Polypill
Number analyzed (Participants) | 153 | 138
mm Hg | 133 (19) | 128 (19)

5. Secondary Outcome: Medication Adherence
Description: polypill-percentage of pills taken, evaluated via pill counts
Time Frame: 2 months
Population: adherence not assessed in usual care arm; incomplete data for 32 polypill participants, resulting in 106 analyzed of 138 polypill participants who completed 2 month visits
Measure: Median (Inter-Quartile Range); unit: percentage of pills taken
Arm/Group | Usual Care | Polypill
Number analyzed (Participants) | 0 | 106
percentage of pills taken |  | 98 [91 to 100]

6. Secondary Outcome: Drug Metabolite Profile
Description: LC/MS/MS-based drug metabolite profile assay screen in the polypill arm.
Time Frame: 12 months
Population: Funding is no longer available to complete the analysis of biomarker measurements. In addition, no future funding is anticipated in order to complete this analysis.
Arm/Group | Usual Care | Polypill
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: LDL Cholesterol
Description: polypill versus usual care
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Usual Care | Polypill
Number analyzed (Participants) | 153 | 137
mg/dL | 108 (35) | 90 (33)

8. Secondary Outcome: Insulin Resistance
Description: Measurement of HOMA-IR using fasting glucose and insulin.
Time Frame: Baseline and 12 months
Population: as for outcome 6
Arm/Group | Usual Care | Polypill
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Inflammatory Profile
Description: Plasma levels of IL-17, IFN-g, IL-6, IL-10, high sensitivity C-reactive protein, TNFa, IL-4.
Time Frame: Baseline and 12 months
Population: as for outcome 6
Arm/Group | Usual Care | Polypill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: For the duration of the study period (Dec 2015 through June 2018) and for each participant's 12-month period of participation
Arm/Group | Usual Care | Polypill
All-Cause Mortality (participants affected / at risk) | 2/155 | 2/148
Serious Adverse Events (participants affected / at risk) | 3/155 | 2/148
Other Adverse Events (participants affected / at risk) | 0/155 | 0/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=155) | Polypill (N=148)
non-CV death (Renal and urinary disorders) | 0 (0) | 1 (1)
non-CV death (Hepatobiliary disorders) | 0 (0) | 1 (1) — alcohol toxicity
stroke-related death (Vascular disorders) | 1 (1) | 0 (0)
death from motor vehicle accident (Social circumstances) | 1 (1) | 0 (0)
Coronary Artery Bypass Surgery (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT02278471/Prot_SAP_000.pdf